CLINICAL TRIAL: NCT01551004
Title: Randomized, Double-Blind, Placebo-Controlled, Single Ascending Dose Phase I Trial to Determine the Safety and Pharmacokinetics of CRS3123 Administered Orally to Healthy Adults
Brief Title: Phase I Trial of a Single Dose of CRS3123
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: National Institute of Allergy and Infectious Diseases (NIAID) (NIH)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Treatment
Other Study IDs: 10-0008; HHSN272201500007I
Record Dates: First submitted 2012-03-08; First posted 2012-03-12 (Estimated); Last update posted 2017-09-25 (Actual); Status verified 2014-09-26

CONDITIONS: Clostridium Difficile Colitis
Keywords: C. diff; C. difficile; Clostridium difficile; CRS3123
MeSH Terms: conditions — Enterocolitis, Pseudomembranous | interventions — REP 3123

STUDY DESIGN:
Who Masked: Participant, Investigator
Oversight: FDA-regulated Drug: Yes | FDA-regulated Device: No | US Export: No

ARMS (5):
- Cohort A (Experimental): 8 subjects (6 active, 2 placebo) receive a single oral dose of 100 mg CRS3123 or placebo
  Interventions: Drug: CRS3123; Other: Placebo
- Cohort B (Experimental): 8 subjects (6 active, 2 placebo) receive a single oral dose of 200 mg CRS3123 or placebo
  Interventions: Drug: CRS3123; Other: Placebo
- Cohort C (Experimental): 8 subjects (6 active, 2 placebo) receive a single oral dose of 400 mg CRS3123 or placebo
  Interventions: Drug: CRS3123; Other: Placebo
- Cohort D (Experimental): 8 subjects (6 active, 2 placebo) receive a single oral dose of 800 mg CRS3123 or placebo
  Interventions: Drug: CRS3123; Other: Placebo
- Cohort E (Experimental): 8 subjects (6 active, 2 placebo) receive a single oral dose of 1200 mg CRS3123 or placebo
  Interventions: Drug: CRS3123; Other: Placebo

INTERVENTIONS:
Drug: CRS3123 — CRS3123, a methionyl-tRNA synthetase inhibitor, will be supplied in 100 and 200 milligram capsules. Subjects randomized to active drug in Cohorts A through E will receive 100 mg, 200 mg, 400 mg, 800 mg and 1200 mg respectively, as a single oral dose.
Other: Placebo — Matching placebo capsules will be given to 2 subjects of each cohort.

SUMMARY:
Double-blind, randomized, placebo-controlled Phase I Trial to determine the safety and pharmokinetics of a single dose of CRS3123 in healthy adult volunteers. Forty healthy male and female subjects 18 to 45 years will be admitted in 5 dosing Cohorts, 8 subjects per Cohort. Up to two alternates may be used per dosing Cohorts for study subjects that drop out. The primary objective of the study is to determine the safety and tolerability of escalating doses of CRS3123 following oral administration to healthy subjects.

DETAILED DESCRIPTION:
This is a Phase I, multi-center, placebo-controlled, double-blind, dose-escalation study to evaluate the safety and tolerability of CRS3123, a methionyl-tRNA synthetase inhibitor. Since this is a FIH study of a new class of drugs, the maximum safe starting dose was estimated from the NOAEL from preclinical studies in accordance with FDA guidance documents (FDA Guidance for Industry, July 2005). A very low starting dose has been chosen. In the initial Cohorts, doses of 100, 200 and 400 will be given; all are below the estimated human starting dose. If any significant safety signals are encountered, the investigators will notify the SMC and call for a review. Dose escalation to Cohorts D and E will require a full SMC review of all safety data obtained through Day 7 for the preceding Cohorts. Forty healthy male and female subjects 18 to 45 years, inclusive, will be admitted for an inpatient study. Each subject will receive a single oral dose of CRS3123 or placebo. There will be 8 patients for each cohort (6 active, 2 placebo). The ascending doses are 100, 200, 400, 800 and 1200 mg respectively for cohorts A through E. The primary objective is the safety and tolerability of escalating doses of CRS3123 following oral administration to healthy subjects. The secondary objective is to assess whether there is measurable systemic exposure and if so, to determine the plasma pharmacokinetic characteristics of CRS3123 after a single oral dose.

ELIGIBILITY:
Inclusion Criteria:

-Men and women 18 to 45 years of age, inclusive -Ability to understand the consent process and procedures -Informed consent obtained and signed -Comprehension of the protocol, which will be determined by the recruiter using a series of questions after explaining the procedures. Spanish speaking subjects will utilize a Spanish translation of the consent form with verbal discussion of the study's consent form and protocol by a JHU certified Spanish interpreter. -Subjects agree to be available for all study visits. Subjects will be asked if they have any travel plans, and whether staff could use alternate contact information that will be provided. -General good health, without current medical illness or clinically significant abnormal physical examination findings that classify the subject as other than healthy as determined by study investigators -Negative serum pregnancy test at screening and a negative urine pregnancy test on the day of admittance to the inpatient phase for all female subjects of child bearing potential -Negative urine toxicity screen for marijuana, cocaine metabolite, amphetamines, opiates, PCP, barbiturates, benzodiazepines -Negative breathalyzer -Body mass index (BMI) of < 35 [weight (kg)]/[height (m)^2] -Agreement by subjects with reproductive potential to use an adequate method of contraception during the study and for 4 weeks after study drug administration. Female subjects must agree to the use of TWO reliable methods of contraception while receiving study drug and for 4 weeks after study drug administration, which can include: condoms, spermicidal gel, diaphragm, hormonal or non-hormonal intrauterine device, surgical sterilization, oral contraceptive pill, depot progesterone injections, and sexual abstinence. If a male subject is sexually active, the subject and his partner mus agree to use at least one of the above listed contraceptive methods. -If the subject uses abstinence and becomes sexually active during the study, they must agree to use TWO if female and one if male, of the above listed contraceptive methods.

Exclusion Criteria:

-Medical condition that precludes participation, including the following: a. Hypertension with confirmed systolic blood pressure >140 mmHg or confirmed diastolic blood pressure >90 mmHg, measured after 10 - 15 minutes of rest b. Morbid obesity (BMI>35) c. Current diagnosis of pulmonary disease d. Current diagnosis of asthma, which has required use of asthma medications within the past year e. History of or current diagnosis of diabetes f. Autoimmune disorder, such as lupus, Wegener's, rheumatoid arthritis g. History of malignancy except low-grade skin cancer, (i.e., basal cell carcinoma has been surgically cured) h. Chronic renal, hepatic, or pulmonary disease condition that could interfere with the absorption of the study drug (e.g., surgical resection of significant proportions of the stomach or bowel, gastric bypass, gastric banding, irritable bowel syndrome, inflammatory bowel disease) i. History of known Clostridium difficile infection j. Blood donation within the previous 6 weeks k. History of cardiac rhythm abnormality including Wolff/Parkinson/White syndrome l. History of prolonged QT interval m. History of ovarian cysts -Prolongation of QTcB interval (i.e., confirmed QTcB interval >450 milliseconds) -Clinically significant abnormal electrocardiogram at screening in the judgment of the investigator, or based on the formal ECG reading; history of any cardiac abnormalities, including conduction abnormalities such as Wolff-Parkinson-White, dysrhythmias, or coronary artery disease -Laboratory values outside the expanded ranges in Appendix B for the following tests: blood cell counts (white blood cell counts [WBC], hemoglobin, platelets), serum chemistry (sodium, potassium, calcium, chloride, CO2, creatinine, glucose, BUN, AST, AP, ALT, total bilirubin, protein, albumin, amylase), urinalysis for glucose, protein and blood(with proviso for re-testing females in Section 6). If CK is above normal range at baseline, but not clinically significant, the subject can be included. -Positive serology results for HIV, HBsAg, or HCV antibodies -Febrile illness with temperature documented >38 degrees C within 7 days of dosing -Pregnancy or breastfeeding -Known allergic reactions to study drug components, including ingredients present in the formulation. -Treatment with another investigational drug within 30 days of dosing -Lack of ability to fully understand the informed consent. This will be determined by the recruiter/interviewer after explaining the consent and observing the subject reading the consent. -Ingestion of prescription medications, grapefruit juice, or St John's Wort starting 14 days or 5 half-lives before dosing, whichever is longer. Women may use oral contraceptives. -Ingestion of herbal supplements or over-the-counter medications starting 7 days before dosing -Use of any form of tobacco, including cigarette smoking, pipe smoking, or oral tobacco; if a former smoker or tobacco user, the subject must not have used tobacco for 30 days before screening -Any specific condition that, in the judgment of the Investigator, precludes participation because it could affect subject safety

Ages: 18 Years to 45 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult
Enrollment: 40 (Actual)
Dates: Start 2012-05-22 (Actual); Primary Completion 2014-04-07 (Actual); Study Completion 2014-04-21 (Actual)

PRIMARY OUTCOMES:
Changes from baseline in findings on physical examination. | Day 0 to Day 28
Changes from baseline in key ECG findings. | Day 0 to Day 28
Changes from baseline in safety laboratory tests (hematology, chemistry, urinalysis). | Day 0 to Day 28
Changes from baseline in vital sign measurements. | Day 0 to Day 28
Reported adverse events | Day 0 to Day 28

SECONDARY OUTCOMES:
Pharmacokinetics of CRS3123 determined and compared by measuring plasma CRS3123 concentrations before oral administration of CRS3123 and at multiple specified time points following dose administration. | Day 0 Pre-dose and at the following times after dosing: 15 and 30 minutes, and 1, 2, 3, 4, 6, 8, 10, 12, 24, 48, and 72 hrs.
Pharmacokinetics of CRS3123 determined and compared by measuring urine CRS3123 concentrations before oral administration of CRS3123 and at multiple specified time points following dose administration. | Day 0, 24 hour timed urine collection after dosing.

CONTACTS AND LOCATIONS:
Locations (1):
- Johns Hopkins Bayview Medical Center - Infectious Diseases, Baltimore, Maryland, United States

REFERENCES:
- [Derived] Nayak SU, Griffiss JM, Blumer J, O'Riordan MA, Gray W, McKenzie R, Jurao RA, An AT, Le M, Bell SJ, Ochsner UA, Jarvis TC, Janjic N, Zenilman JM. Safety, Tolerability, Systemic Exposure, and Metabolism of CRS3123, a Methionyl-tRNA Synthetase Inhibitor Developed for Treatment of Clostridium difficile, in a Phase 1 Study. Antimicrob Agents Chemother. 2017 Jul 25;61(8):e02760-16. doi: 10.1128/AAC.02760-16. Print 2017 Aug. PMID 28584140